CLINICAL TRIAL: NCT02986594
Title: Shanghai First Maternity and Infant Hospital, Tongji University School of Medicine
Brief Title: Diagnosis and Treatment Strategy of Recurrent Spontaneous Abortion Associated With Thrombophilla
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Shihua Bao, Principal Investigator, Shanghai First Maternity and Infant Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiFIMH-0002
Record Dates: First submitted 2016-11-27; First posted 2016-12-08 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-11

CONDITIONS: Thrombophilia With Recurrent Pregnancy Loss
MeSH Terms: interventions — Aspirin; Heparin

ARMS (3):
- aspirin group (Experimental): low dose aspirin, 75-100mg, bid, after pregnancy
  Interventions: Drug: Aspirin
- low molecular weight heparin group (Experimental): low molecular weight heparin, 4100u, qd, after pregnancy
  Interventions: Drug: Heparin
- combination group (Experimental): low molecular weight heparin, 4100u, once a day and low dose aspirin, 75-100mg, bid. After pregnancy
  Interventions: Drug: Aspirin; Drug: Heparin

INTERVENTIONS:
Drug: Aspirin
  Arms: aspirin group; combination group
Drug: Heparin
  Arms: combination group; low molecular weight heparin group

SUMMARY:
In this clinical cohort study, the investigators observe the efficacy of low molecular weight heparin in the treatment of thrombophilia with recurrent pregnancy loss with a prospective randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Woman who had their Second miscarriage before 12(th) week of gestation.The patient who is diagnosed as thrombophilia with recurrent pregnancy loss. Signed consent form.

Exclusion Criteria:

1. having experiencedsevere allergies, trauma history and/or operation history within 3 months
2. with a history of mental illness and/or family history of mental illness
3. limb disabled
4. taking medicine within one month
5. suffering major events or having mood swings
6. with a history of recurrent pregnancy loss
7. having internal and surgical disease(after having variety of physical examination such as electrocardiogram/hepatic and renal function/blood routine and urine rotine)
8. Chromosome aberrations in anyone of the couple.
9. patients who have drug contraindications

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
D-Dimer | through study completion, an average of 3 year

SECONDARY OUTCOMES:
BMI in kg/m^2 | through study completion, an average of 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai first Maternity and Infant health hospital, Tong Ji University, Shanghai, China